CLINICAL TRIAL: NCT03095872
Title: Comparison of the Effect of Vaseline and Bepanthen® "Wund- Und Heilsalbe" on the Wound Healing Following Fractional Ablative Laser Treatment of Photo-damaged Skin
Brief Title: Comparison of the Effect of Vaseline and Bepanthen® "Wund- Und Heilsalbe" on the Wound Healing Following Laser Therapy
Acronym: CO2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-011
Record Dates: First submitted 2017-02-24; First posted 2017-03-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Photodamaged Skin
Keywords: photodamaged skin; wound healing; CO2 laser
MeSH Terms: interventions — Lasers, Gas; Petrolatum; dexpanthenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bepanthen/Vaseline (Experimental): One half of the wound occuring after CO2 laser therapy of photo-damaged skin is treated with Bepanthen and the other half with Vaseline.
  Interventions: Device: CO2-laser; Drug: Vaseline; Drug: Bepanthen

INTERVENTIONS:
Device: CO2-laser — Patients with photo-damaged skin are treated with the CO2 laser to remove damaged skin layers.
Drug: Vaseline — After the laser treatment, the wound area will be divided into two parts with a sterile skin marker. One area will be treated with Vaseline, and be marked "V". Thus, it is ensured that the care product will be applied correctly to the defined area. Postoperatively, this area of the wound will be treated with Vaseline. In the next seven days the patient will repeat the treatment every day at home.
Drug: Bepanthen — After the laser treatment, the wound area will be divided into two parts with a sterile skin marker. One area will be treated with Bepanthen® Wund- und Heilsalbe, and be marked "B". Thus, it is ensured that the care product will be applied correctly to the defined area. Postoperatively, this area of the wound will be treated with Bepanthen® Wund- und Heilsalbe. In the next seven days the patient will repeat the treatment every day at home.

SUMMARY:
In the field of dermatology the healing process and therefore the success of a laser treatment are strongly determined by an appropriate postoperative treatment of the laser-treated skin. The manufacturer of CO2 laser systems recommends the application of Vaseline postoperatively to protect the treated tissue from air exposition until encrustation of the laser-treated skin decreases (usually after 7-14 days). An alternative to Vaseline could be Bepanthen® "Wund- und Heilsalbe" (Bayer). It contains the active ingredient pro-vitamin Dexapanthenol, which is widely used in dermatology therapy. The product helps to stabilize the protective barrier of the skin, to reduce the skin irritation, to stimulate the skin regeneration and to promote the wound healing. In an in-vitro study Bepanthen® "Wund- und Heilsalbe" triggered wound closure significantly faster compared to Vaseline. In this study the effect of Bepanthen® "Wund- und Heilsalbe" on wound healing should be investigated and compared to Vaseline in vivo following fractional ablative CO2 laser treatment of photo-damaged skin.

DETAILED DESCRIPTION:
The healing process and therefore the success of a laser treatment are strongly determined by an appropriate treatment with special skin care products of the laser-treated skin. Cooling measures prevent the swelling of the treated skin area, if applied directly after the procedure. A soothing and wound-healing-promoting care applied subsequently for seven days, can support and also speed up the healing process.

The Lumenis® Company is the manufacturer of CO2 laser systems and recommends the application of the Okklusiv ointment Vaseline® postoperatively, in order to prevent the treated tissue to the air exposition. These occlusive wound care should be maintained, until the encrustation of the laser-treated skin decreases, which usually happens 7-14 days postoperatively.

The Bepanthen® Wund- und Heilsalbe (Bayer) could be a possible alternative to Vaseline® as postoperative care. Bepanthen® Wund- und Heilsalbe contains pro-vitamin Dexpanthenol as an active ingredient and is widely used in dermatological therapy. The product helps to stabilize the protective barrier of the skin, to reduce the skin irritation, to stimulate the skin regeneration and to promote the wound healing. The investigators examined the effect of substances containing Dexpanthenol on wound healing process applied topically, in three-dimensional (3D) dermal skin equivalents in vitro. For this purpose, many lesions with standardized diameter and depth were generated using a laser. The subsequent topical application of substances containing dexpanthenol on the wound healing models (treated with laser) for three-days led to a significantly faster wound closure compared to Vaseline-covered models (Marquardt et al., 2015). The aim of this study is to compare the effect of white Vaseline with Bepanthen® "Wund- und Heilsalbe" (both applied postoperatively) on the wound healing following fractional ablative CO2 laser treatment of photo-damaged skin in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* photodamaged skin, which need to be treated with the fractional ablative CO2 laser

Exclusion Criteria:

* pregnant or lactating females
* chronic diseases such as diabetes and vascular disease with impaired wound healing
* Patients, who tend to form hypertrophic scars and keloids
* Patients, who take the isotretinoin-containing medication in the past year
* topical or systemic corticosteroid treatment
* immunocompromised patients
* Patients with the Koebner phenomenon
* People with the skin type 6
* Patients with melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
Change of the diameter of the individual lesions [initial value 1.3mm] between study visits. | Over 2 weeks (immediately after laser treatment and on day 1, 2, 5 and 14 after laser treatment)
  Large clinical digital photos as well as dermatoscopic images of the skin.
Change of the size of the individual lesions between study visits. | Over 2 weeks (immediately after laser treatment and on day 1, 2, 5 and 14 after laser treatment)
  Two-dimensional microscopic skin cut images in real time of the skin.
Visual changes of the wound healing between study visits. | Over 2 weeks (immediately after laser treatment and on day 1, 2, 5 and 14 after laser treatment)
  The wound healing rates will be visually assessed, based on the measure of re-epithelialization.
Change of the wound under cosmetic aspects between study visits. | Over 2 weeks (immediately after laser treatment and on day 1, 2, 5 and 14 after laser treatment)
  The cosmetic result is based on a visual analog scale (VAS) from 0 (bad) to 10 (excellent, with no visible difference of the wound to the surrounding tissue).

SECONDARY OUTCOMES:
Change of the transepidermal water loss (TEWL) between study visits. | Over 2 weeks (immediately after laser treatment and on day 1, 2, 5 and 14 after laser treatment)
  TEWL is the most important parameter for the assessment of skin barrier function.

CONTACTS AND LOCATIONS:
Overall Officials: Jens M. Baron, Prof. Dr. med., Principal Investigator — RWTH Aachen University, Department of Dermatology and Allergology
Locations (1):
- University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bogdan Allemann I, Kaufman J. Laser principles. Curr Probl Dermatol. 2011;42:7-23. doi: 10.1159/000328236. Epub 2011 Aug 16. PMID 21865794
- [Background] Reinholz M, Tietze JK, Kilian K, Schaller M, Schofer H, Lehmann P, Zierhut M, Klovekorn W, Ruzicka T, Schauber J. Rosacea - S1 guideline. J Dtsch Dermatol Ges. 2013 Aug;11(8):768-80; 768-79. doi: 10.1111/ddg.12101. Epub 2013 May 6. No abstract available. English, German. PMID 23647643
- [Background] Marquardt Y, Amann PM, Heise R, Czaja K, Steiner T, Merk HF, Skazik-Voogt C, Baron JM. Characterization of a novel standardized human three-dimensional skin wound healing model using non-sequential fractional ultrapulsed CO2 laser treatments. Lasers Surg Med. 2015 Mar;47(3):257-65. doi: 10.1002/lsm.22341. Epub 2015 Mar 15. PMID 25771913
- [Background] Wigger-Alberti W, Kuhlmann M, Ekanayake S, Wilhelm D. Using a novel wound model to investigate the healing properties of products for superficial wounds. J Wound Care. 2009 Mar;18(3):123-28, 131. doi: 10.12968/jowc.2009.18.3.39813. PMID 19247233
- See also: Leitlinie zur Behandlung der aktinischen Keratosen C44.X der Deutschen Dermatologischen Gesellschaft. — http://www.escf-network.eu/fileadmin/user_upload/Files/Leitlinie_AK_K5_Ds.pdf